CLINICAL TRIAL: NCT05628116
Title: Double-blind, Randomized, Placebo-controlled, Phase I Clinical Study of the Safety, Tolerability and Pharmacokinetics of Ascending Doses of X243 After Single and Multiple Oral Administration in Healthy Volunteers.
Brief Title: Double-blind, Randomized, Placebo-controlled Study of the Safety, Tolerability and Pharmacokinetics of Ascending Doses of XC243 After Single and Multiple Oral Administration in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PHARMENTERPRISES LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PAIN-ХС243-01
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteers
Keywords: Phase 1
MeSH Terms: interventions — Single Person

STUDY DESIGN:
Intervention Model Description: The dose cohorts will be included into the study subsequently based on preliminary safety results evaluation performed by the DSMC. 2 doses of XC243/placebo (50 mg, 100 mg) were used in the single-dose ascending study. 1 dose of XC243/placebo (200 mg) were used in the single-dose food effect study. 1 dose of XC243/placebo (200 mg) were used in the repeated dose study.The duration of exposure to the ID is planned 1 day in single dosing cohorts and 14 days in multiple dosing cohort.
Who Masked: Participant, Investigator
Masking Description: Blinding was carried out by using placebo equivalent to XC243 tablets without active pharmaceutical ingredients (API) and the corresponding labeling of the ID.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- XC243 50 mg single (Experimental): Cohort 1 - 7 subjects will be randomized in a 5:2 ratio to be treated either XC243 50 mg (5 subjects) or placebo (2 subjects, see placebo single arm)
  Interventions: Drug: XC243 50 mg single
- XC243 100 mg single (Experimental): Cohort 2 - 7 subjects will be randomized in a 5:2 ratio to be treated either XC243 100 mg (5 subjects) or placebo (2 subjects, see placebo single arm)
  Interventions: Drug: XC243 100 mg single
- Placebo single (Placebo Comparator): Placebo comparator arm will consist of 4 subjects (1 subject each from Сohorts 1 and 2)
  Interventions: Drug: Placebo single
- XC243 200 mg single-dose food effect (Experimental): Cohort 3 - 14 subjects will be randomized in a 12:2 ratio to be treated either XC243 200 mg (12 subjects) or placebo (2 subjects, see placebo single arm) first on an empty stomach, and after the washing period after eating
  Interventions: Drug: XC243 200 mg single-dose food effect
- Placebo single-dose food effect (Placebo Comparator): Placebo comparator arm will consist of 2 subjects from Cohort 3
  Interventions: Drug: Placebo single-dose food effect
- XC243 200 mg multiple (Experimental): Cohort 4 - 10 subjects will be randomized in a 8:2 ratio to be treated either XC243 200 mg (8 subjects) or placebo (2 subjects, see placebo multiple arm)
  Interventions: Drug: XC243 200 mg multiple
- Placebo multiple (Placebo Comparator): Placebo comparator arm will consist of 2 subjects from cohort 4
  Interventions: Drug: Placebo multiple

INTERVENTIONS:
Drug: XC243 50 mg single — The volunteers will receive a single dose of the ID (1 tablet once, 50 mg)
  Arms: XC243 50 mg single
Drug: XC243 100 mg single — The volunteers will receive a single dose of the ID (2 tablets once, 100 mg)
  Arms: XC243 100 mg single
Drug: Placebo single — The volunteers will receive a single dose of the ID (1 or 2 tablets once)
  Arms: Placebo single
Drug: XC243 200 mg single-dose food effect — The volunteers will receive single dose of the ID during first on an empty stomach, and after the washing period after eating (4 tablets, 200 mg)
  Arms: XC243 200 mg single-dose food effect
Drug: Placebo single-dose food effect — The volunteers will receive single dose of the ID during first on an empty stomach, and after the washing period after eating (4 tablets)
  Arms: Placebo single-dose food effect
Drug: XC243 200 mg multiple — The volunteers will receive multiple doses of the ID during 14 days (4 tablets daily, 200 mg each)
  Arms: XC243 200 mg multiple
Drug: Placebo multiple — The volunteers will receive multiple doses of the ID during 14 days (4 tablets daily)
  Arms: Placebo multiple

SUMMARY:
A double-blind, randomized, placebo-controlled, Phase I clinical study of the safety, tolerability and pharmacokinetics (PK) of ascending doses of XC243 after single and multiple oral administration in healthy volunteers. It's planned to include sequentially 2 cohorts of 7 volunteers who will receive a single dose of XC243 (50 mg and 100 mg) or placebo (cohort ratio 5:2), 1 cohort of 14 volunteers who will receive a single dose of XC243 200 mg or placebo first on an empty stomach, and after the washing period after eating (cohort ratio 12:2) and 1 cohort of 10 volunteers who will receive XC243 200 mg or placebo on an empty stomach during 14 days (cohort ratio 8:2).

DETAILED DESCRIPTION:
The study will be conducted in 1 centre. The study will consist of 3 parts: single-dose ascending study, single-dose food effect study for dose 200 mg, repeated dose study of 200 mg over 14 days.

The volunteers of single dosing cohorts will receive the investigated drug (ID) ХС243 or placebo once and stay at the study center for at least 24 hours after the ID administration to monitor the safety parameters and for sampling for PK analysis. The Follow-up will last 7 days, during which safety parameters and PK in volunteers will be studied. Based on all safety data from the XC243 50 mg cohort, the Data Safety Monitoring Committee (DSMC) will consider dose increase and entry of the 100 mg cohort. If the single dose of ХС243 100 mg is considered to be safe, the third dosing cohort of 200 mg will be included in the single-dose food effect study.

The volunteers of third dosing cohort will receive the ID ХС243 (200 mg) or placebo once on an empty stomach.The Follow-up will last 7 days, during which safety parameters and PK in volunteers will be studied. The washing period will last 7 days, after which volunteers will receive the ID ХС243 (200 mg) or placebo once after eating. The Follow-up will last 7 days too. If the single dose of ХС243 200 mg is considered to be safe, the fourth multiple dosing cohort of repeated dose of 200 mg will be included.

The volunteers from multiple dosing cohort will receive the ID (ХС243 or placebo) once a day during 14 days and will stay at the hospital (study center) within 15 days. The Follow-up will last 14 days, during which they will study safety parameters and PK in volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. The volunteer read, understood and signed the Information Leaflet and the Informed Consent Form to participate in the study;
2. Non-smoking men (nonsmokers at least within the last year before the screening) at the ages from 18 through 45;
3. Verified diagnosis "healthy" according to standard clinical, laboratory and instrumental methods of examination;
4. Blood Pressure (BP): Systolic blood pressure (SBP) 100 to 130 mm Hg, diastolic blood pressure (DBP) from 70 to 89 mm Hg (inclusive);
5. Heart rate (HR) from 60 to 90 units/min (inclusive);
6. Respiratory rate (RR) from 12 to 20 min-1 (inclusive);
7. Body temperature from 36 to 36.9 ° C (inclusive);
8. Body mass index from 18.5 to 30.0 kg/m2 with body weight of more than 45 kg and no more than 110 kg;
9. Negative result of breath alcohol test, urine test for narcotic substances;
10. Consent to use adequate contraceptive methods throughout the study, including the post-observation period (7 days in Cohorts 1-3 and 14 days in Cohort 4), as well as 90 days at its end;
11. Agreement to observe the daily and nutritional regimen provided for by the study protocol.

Exclusion Criteria:

1. The history of chronic diseases of the cardiovascular, bronchopulmonary, nervous, endocrine, musculoskeletal system, as well as the gastrointestinal tract (GI), liver, kidneys, blood, mental illness, epilepsy or seizure;
2. Deviations of standard laboratory and instrumental values, as well as physical examination results from normal values at screening;
3. History of GI surgery (excluding appendectomy);
4. Administration of drugs less than 2 weeks before screening (including preparations of plant origin, vitamins and dietary supplements), with the exception of episodic administration of paracetamol at a dose of up to 1.5 g/day;
5. Taking drugs that affect liver function (for example, inhibitors and/or inducers of cytochrome P450) less than 30 days before screening;
6. Presence of antibodies to HIV and hepatitis C virus at screening, presence of hepatitis B virus surface antigen, presence of antibodies to T. Pallidum *;
7. Presence of a positive test for SARS-CoV-2 at screening;
8. Presence of unstable sleep structure (for example, night shift work, sleep disturbances, insomnia, recent return from another time zone, etc.), extreme physical activity (for example, lifting weights);
9. A special diet (for example, vegetarian, vegan, hypocaloric (less than 1000 kcal/day));
10. Taking alcohol within 4 days of screening or testing positive for exhaled alcohol at screening or on Day -1;
11. Taking narcotic drugs within 4 days before screening or a positive urine drug test at screening or on Day -1;
12. History of alcohol and/or drug dependence or intake of more than 5 units of alcohol per week (one unit of alcohol is 40 ml of strong alcoholic beverages, 330 ml of beer or 150 ml of wine) since the beginning of the screening stage;
13. Smoking or using nicotine-containing products at present and for 6 months prior to screening;
14. History of allergic and/or hypersensitivity reactions to drugs;
15. Hypersensitivity to study drug components;
16. Blood/plasma donation (450 ml blood or plasma or more) less than 2 months prior to screening;
17. Vaccination with live vaccines less than 90 days before screening;
18. Participate in other clinical trials or take study medication within 3 months prior to screening. Volunteers who have not been screened in another study, as well as volunteers who have not been included in another study, can be included in this study;
19. Acute infectious diseases less than 4 weeks prior to screening;
20. Inability to read or write; unwillingness to understand and follow study protocol procedures; failure to perform procedures that the Investigator believes may affect the study results or safety of the volunteer and prevent the volunteer from entering the study;
21. Any concomitant medical or serious mental conditions that render a volunteer unfit to participate in a clinical trial limit the validity of obtaining informed consent or may affect the volunteer's ability to participate in the study, in the reasonable opinion of the study physician;
22. Site staff, regardless of participation in this clinical trial, members of their families or subjects in dependent relationships.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events (AEs) per treatment arm | Day 1-Day 35
  Adverse events will be classified according to CTCAE. Adverse events will be summarized descriptively by treatment arm. Verbatim terms will be mapped to preferred terms and organ systems using the current Medical Dictionary for Regulatory Activities version.

SECONDARY OUTCOMES:
Pharmacokinetics of XC243 by assessing AUC0-inf | Day 1- Day 14
  Area under the curve "concentration of the drug-time" from the time of administration of the drug till infinity.
Pharmacokinetics of XC243 by assessing Cmax | Day 1- Day 14
  Maximum plasma concentration
Pharmacokinetics of XC243 by assessing AUC0-t | Day 1- Day 14
  Area under the curve "concentration of the drug-time" from the time of administration of the drug till the time (t) the last blood sampling
Pharmacokinetics of XC243 by assessing Tmax | Day 1- Day 14
  Time to maximum drug concentration in the blood plasma administration
Pharmacokinetics of XC243 by assessing T1/2 | Day 1- Day 14
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Locations (1):
- LLS X7 Clinical Research, Saint Petersburg, Russia